CLINICAL TRIAL: NCT04565743
Title: Stop At One Stockholm: Co-operation Between Health Care Providers and Medical Education in Primary Health Care to Prevent Falls and Fractures in the Elderly
Brief Title: Stop At One Stockholm (SAOS)- Secondary Fracture Prevention Through Active Patient Identification and Staff Education.
Acronym: SAOS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Helena Salminen (Other)
Collaborators: Region Stockholm (Other Government)
Responsible Party: Sponsor-Investigator, Helena Salminen, Associate professor, Karolinska Institutet
Organization: Karolinska Institutet (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2018/927-31/2
Record Dates: First submitted 2020-09-17; First posted 2020-09-25 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2024-04

CONDITIONS: Osteoporotic Fractures; Osteoporosis; Osteoporosis Risk
Keywords: Organization & administration; Secondary prevention; Bone Density Conservation Agents
MeSH Terms: conditions — Osteoporotic Fractures; Osteoporosis

STUDY DESIGN:
Intervention Model Description: Cluster randomized controlled study. 40 clusters with an estimated cluster size of 90 participating individuals in each cluster.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Active Comparator): Multiprofessional education for health professionals in primary care on secondary prevention of osteoporotic fractures. Identification and referral of patients with recent osteoporotic fracture.
  Interventions: Behavioral: Support on dentification and treatment of patients with high risk of osteoporotic fractures
- Control (No Intervention): No intervention from study. No restrictions regarding education or the local organization of care for the prevention of osteoporotic fractures.

INTERVENTIONS:
Behavioral: Support on dentification and treatment of patients with high risk of osteoporotic fractures — Education for primary care health care professionals and referral of patients with recent osteoporotic fracture.
  Arms: Intervention

SUMMARY:
This is a study on the effects of education on secondary fracture prevention in primary health care centers (PHCC) and referral from hospitals to these PHCC of patients with recent fragility fractures.

The design is Cluster-randomized controlled study with two arms. 40 primary health care centers (PHCC) are included, each PHCC constitutes a cluster. The intervention group contains 20 PHCCs and the control group of the remaining 20 PHCCs. The educational part of the intervention is divided into three sessions; one web based course succeeded by two multiprofessional seminars with six months interval. During the intervention period patients enlisted at the intervention PHCCs, aged 60 or more who are diagnosed on a fragility fracture are referred to their respective PHCC. The primary outcome are the proportions of patients who receive bone specific treatment after their fracture in the intervention group compared to the control group.

DETAILED DESCRIPTION:
Fragility fractures are in this study defined as a fracture of the spine, hip, pelvis, proximal humerus och distal radius caused by low energy trauma. A trauma not exceeding the force implied on the body from a fall from standing height on a flat surface, is regarded to be a low energy trauma.

The educational intervention targets general practitioners and nurses from the PHCC as well as physiotherapists, occupational therapists and dietitians from a nearby rehabilitation centre.

All professions go through the same web course before educational session #1 which is held at the PHCC. The web course includes basic knowledge about risk factors for fragility fractures

At session #1 all professions first participate in a common seminar of 45 minutes. After that physicians, nurses and rehabilitation related professions each have an additional seminar of 45 minutes, that means three separate seminars. Three teachers lead the seminars; a specialist in family medicine, a nurse specialized in primary care and a physiotherapist. They are all present during all of the seminars at each PHCC and the same three individuals leads the seminars at all PHCCs. The seminars focus on identification of persons at high risk of fracture and different methods to lower that risk. The importance of multiprofessional care for these patients is stressed. The participants are given opportunity to discuss how they might facilitate cooperation between the different health vare professions. Development of local routines for multiprofessional care is encouraged.

Educational session #2 is held approximally 6 months after session #1. Session #2 invites the same health care professionals as session #1. There are three parts. A first part of 45 minutes for the physicians and nurses. A second part of 45 minutes where personnel from the rehabilitation center joins. The third part of 45 minutes includes just the rehabilitation personnel.

At session #2 includes a short review of the contents discussed in session #1. The focus however is on the development of new local routines to secure the ability for patients with a high risk of fracture to be offered multiprofessional care. What needs to be done and who does what at your PHCC/rehabilitation center? The participants also get feedback on the number of patients being treated with bone-specific drugs before and after the start of the intervention.

Inclusion of patients stops at december 1 2020. Referrals to the PHCC of the patients included last will be conducted during January 2021.

Primary outcome data is gathered at each PHCC from the medical journals of the enlisted patients aged >60 with fragility fractures. Data includes the time frame one year before start of study, until two years after the last patient was included.

Secondary outcomes, fractures and fall related injuries will be collected from National health care registers, three and five years after the last patient was included.

ELIGIBILITY:
All primary health care centers (PHCCs) in Stockholm County were invited to participate in the study. The goal was to include at least 40

Inclusion Criteria for referral of patients to PHCC:

* Patient has a diagnose at a medical care unit within Stockholm county on a low energy fracture of hip, pelvis, spine, proximal humerus och distal radius between three months before study start an end of study.
* Patient is enlisted at one of the PHCCs in the interventional arm of the study
* Patent is aged 60 years or older

Exclusion Criteria:

* The patient has after the index fracture, already been referred to the correct primary health care center for secondary fracture prevention.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3600 (Estimated)
Dates: Start 2018-02-01 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants treated with bone specific drugs after first fragility fracture at different points in time up to three years after inclusion. | Three years after inclusion of study participant
  Participants are included in the study at the date of their first fragility fracture within the study period. The proportion of participants treated with bone-specific drugs any time since the fracture date, will be measured every 6 months during the study period.

SECONDARY OUTCOMES:
Proportion of participants treated with calcium and vitamin D but not bone specific drugs after first fragility fracture at different points in time after inclusion up to three years after inclusion. | Three years
  Participants are included in the study at the date of their first fragility fracture within the study period. The proportion of participants treated with Calcium and vitamin D supplements but not simultaneously with bone-specific drugs at any time since the fracture date, will be measured until three years after inclusion.

OTHER OUTCOMES:
Incidence of new fractures and fall related injuries after index fracture. | Three and sive years after last participant was included,
  Participants are included in the study at the date of their first fragility fracture within the study period. Mortality, fractures and other fall related injuries are collected from National health care registers for the period three and five years after the last patient was included in the study. The follow up time will thus be different for different participants depending on the date of inclusion.

CONTACTS AND LOCATIONS:
Overall Officials: Helena Salminen, MD, Ass Prof, Principal Investigator — Karolinska Institutet
Locations (1):
- Karolinska Instititet, Huddinge, Stockholm County, Sweden